CLINICAL TRIAL: NCT05730075
Title: The Home-Based Child Care Toolkit for Nurturing School-Age Children Pilot Study
Status: Completed | Type: Observational
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Children's Bureau - Administration for Children and Families (Other); Office of Planning, Research & Evaluation (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 50884
Record Dates: First submitted 2023-01-26; First posted 2023-02-15 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2023-02

CONDITIONS: Child
Keywords: childcare; quality measures; early education; children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Phase 1 HBCC providers: This group will include up to 9 Spanish-speaking HBCC providers, who will receive the Spanish version of the provider questionnaire.
- Phase 1 families: This group will include up to 9 Spanish speaking families and up to 9 English speaking families who will each receive the family questionnaire and who will participate in cognitive interviews.
- 2 HBCC providers: This group will include 150 purposively selected providers from diverse backgrounds who will each complete the provider questionnaire and will also be asked to recruit one or more families to complete the family questionnaire.
- Phase 2 families: This group will include up to 150 purposively selected families who will each receive the family questionnaire.

SUMMARY:
The goal of this observational study is to pilot test the Home-Based Child Care Toolkit for Nurturing School-Age Children (HBCC-NSAC Toolkit) with providers of home-based child care. The main questions it aims to answer are: 1) the extent to which the questionnaires contained in the HBCC-NSAC Toolkit are a reliable and valid measure of HBCC quality and 2) the extent to which the statements and questions in the Toolkit are appropriate for HBCC providers with diverse characteristics and for families who receive care from an HBCC provider. Participants will complete the questionnaires in the Toolkit and participate in cognitive interviews about the questionnaires.

DETAILED DESCRIPTION:
Home-based child care (HBCC), or child care and early education (CCEE) offered in a provider's or child's home, is the most common form of nonparental child care in the United States and is essential for many families. Families of color, those from immigrant backgrounds, those with low incomes who work nontraditional hours, and those living in rural areas are more likely to use HBCC than center-based care.

However, existing quality measures used in HBCC settings are often based on or designed to parallel measures of center-based CCEE. These measures may miss important features of HBCC, such as ways this CCEE meets the needs of families and features that may support positive outcomes for these children and families.

The Home-Based Child Care Supply and Quality (HBCCSQ) project being conducted by Mathematica and Erikson Institute is developing a Home-Based Child Care Toolkit for Nurturing School-Age Children. The toolkit, which contains questionnaires for providers and families, will help HBCC providers who care for at least one school-age child (age 5 and in kindergarten, or ages 6 through 12) in a home setting identify and reflect on their strengths and areas of growth related to their caregiving practices and how they partner with children's families. The purpose of this study is to test the toolkit and ensure its appropriateness for HBCC providers with diverse characteristics and for families who receive care from an HBCC provider.

This pilot study will test the HBCC-NSAC Toolkit in two phases, (1) a pre-test of the Spanish version of the provider questionnaire and the Spanish and English versions of the family questionnaire and (2) a pilot of the full HBCC-NSAC Toolkit (in English and Spanish) and related recruitment and data collection procedures.

In phase one, the study team will recruit up to 9 purposively selected Spanish speaking HBCC providers to complete the Spanish version of the provider questionnaire. Up to 9 Spanish speaking families and up to 9 English speaking families will be purposively selected to complete the family questionnaire. The study team then will conduct a cognitive interview with each provider and family respondent.

In phase two, the study team will recruit 150 purposively selected providers from diverse backgrounds to complete the provider questionnaire. The study team will ask providers to recruit one or more families to complete the family questionnaire on paper, for a total of up to 150 families.

Results from the pilot study will be used to provide initial evidence of the psychometric properties of the items and potentially refine the study instrument for use with a larger number of providers and families in a future validation study.

ELIGIBILITY:
Inclusion criteria:

* Home-based child care providers who care for at least one school-age child (age 5 and in kindergarten, or ages 6 through 12) in a home setting for at least 10 hours per week (within the past year).
* The families must be the primary caregivers of school-age children who receive care in a home-based child care setting for at least 10 hours per week.

Exclusion Criteria:

* Child care providers who do not care for at least one school-age child in a home setting for at least 10 hours per week.
* Primary caregivers (families) who do not have school-age children who receive child care in a home for at least 10 hours per week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consists of home-based child care providers and families who receive child care in a home for at least 10 hours per week.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
The Home-Based Child Care Toolkit for Nurturing School-Age Children | 12 months
  We will assess the validity of the scale by administering the toolkit to HBCCs and families receiving home-based child care.

CONTACTS AND LOCATIONS:
Overall Officials: Sally Atkins-Burnett, Principal Investigator — Mathematica Policy Research, Inc.; Patricia Del Grosso, Study Director — Mathematica Policy Research, Inc.; Ashley Kopack Klein, Study Director — Mathematica Policy Research, Inc.
Locations (1):
- Mathematica Policy Research, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No